CLINICAL TRIAL: NCT00004787
Title: Phase II Pilot Study of Granulocyte Colony-Stimulating Factor for Inherited Bone Marrow Failure Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: James Whitcomb Riley Hospital for Children (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11877; UTMB-416
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Shwachman Syndrome; Fanconi's Anemia; Dyskeratosis Congenita; Thrombocytopenia
Keywords: Fanconi's anemia; Shwachman syndrome; aplastic anemia; dermatologic disorders; dyskeratosis congenita; hematologic disorders; rare disease; thrombocytopenia
MeSH Terms: conditions — Shwachman-Diamond Syndrome; Fanconi Anemia; Dyskeratosis Congenita; Thrombocytopenia; Anemia, Aplastic; Skin Diseases; Hematologic Diseases; Rare Diseases | interventions — Filgrastim

INTERVENTIONS:
Drug: filgrastim

SUMMARY:
OBJECTIVES: I. Assess the efficacy of recombinant human granulocyte colony-stimulating factor (G-CSF) in raising the absolute neutrophil count, platelet count, and hemoglobin level in patients with inherited bone marrow failure syndromes.

II. Assess the efficacy of a reduced maintenance dose in patients who respond to daily G-CSF.

III. Assess the toxic effects of G-CSF in these patients. IV. Measure bone marrow progenitor colonies before and after G-CSF. V. Measure CD34-positive cells in marrow and blood before and after G-CSF using flow cytometry and immunohistochemistry.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive granulocyte colony-stimulating factor (G-CSF) subcutaneously every day for 8 weeks; nonresponders receive an increased dose for an additional 8 weeks. Patients who respond at week 8 or 16 are then tapered to a lower maintenance dose of G-CSF administered every other day through week 40. The dose is adjusted to maintain an absolute neutrophil count above 1500.

Patients are removed from study for failure to achieve a complete response by week 16, unacceptable nonhematologic toxicity, the identification of a clonal karyotype in marrow, or the onset of leukemia.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Inherited bone marrow failure syndrome, including:

* Fanconi's anemia
* Dyskeratosis congenita
* Shwachman syndrome
* Amegakaryocytic thrombocytopenia
* Decreased megakaryocytes in infancy
* No thrombocytopenia with absent radius syndrome (TAR)
* No trisomy 13 or 18
* No clonal bone marrow karyotype

--Prior/Concurrent Therapy--

* At least 4 weeks since growth factors
* Concurrent therapy allowed if not altered for 30 days prior to entry through week 8
* No concurrent investigational drugs

--Patient Characteristics--

* Hematopoietic: ANC <1000
* No leukemia
* Other: No medical or psychiatric contraindication to protocol participation
* No pregnant or nursing women

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1994-12

CONTACTS AND LOCATIONS:
Overall Officials: David A. Williams, Study Chair — James Whitcomb Riley Hospital for Children

REFERENCES:
- [Background] Rackoff WR, Orazi A, Robinson CA, Cooper RJ, Alter BP, Freedman MH, Harris RE, Williams DA. Prolonged administration of granulocyte colony-stimulating factor (filgrastim) to patients with Fanconi anemia: a pilot study. Blood. 1996 Sep 1;88(5):1588-93. PMID 8781414